CLINICAL TRIAL: NCT03819621
Title: Objective Assessment of Orbital Implant and Ocular Prosthesis Motility Using a Digital Imaging
Brief Title: Digital Imaging Assessment of Ocular Prosthesis Motility
Acronym: OCUPEYE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Moorfields Eye Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SAGM1005
Record Dates: First submitted 2018-05-24; First posted 2019-01-28 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Enucleated; Eye
Keywords: Prosthetic; Eye; Enucleation

STUDY DESIGN:
Intervention Model Description: Pilot study to evaluate the mediGrid App against the gold standard rule as a measuring device.
Masking Description: Non-masked study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OCULAR PROSTHESIS MOTILITY (Experimental): All participants ocular prosthesis motility will be measured using the mediGrid app, Image J software in comparison to the ruler as a gold standard.
  Interventions: Device: IRISS Medical Technologies mediGrid app

INTERVENTIONS:
Device: IRISS Medical Technologies mediGrid app — IRISS mediGrid is standalone software, loaded on a mobile electronic platform, which is intended to record and document ophthalmic and other bodily characteristics and to aid in the diagnosis of abnormalities.

SUMMARY:
This study will evaluate the degree of translational movement loss from orbital implant to ocular prosthesis. This will be measured using two software applications - Image J as well as the mediGrid smartphone app in measuring prosthesis motility by comparing it to the ruler as a "gold" standard.

DETAILED DESCRIPTION:
The fit and function of an ocular prosthetic determines the effective motility (movement) within the patient's eye socket. A poor fitting ocular prosthesis will lead to poor motility, patient discomfort and increased mucus discharge, and can risk the integrity of the anterior surface of the implanted orbit. Currently the method to determine best fit of the ocular prosthesis is dependent upon the ocularist's skill in adding or subtracting material from the wax model that is replicated from an initial alginate impression of the patient's eye socket.

The proposal of this study is to utilise digital imaging to capture images to measure the motility of both the orbital implant and the ocular prosthesis. Two methods will be compared: excursion measurements on a photograph using digital software (Image J) versus use of a smart phone app (an iOS app known as mediGrid (IRISS Medical Technologies, UK; CE Marked, HIPAA compliant). This study will evaluate the degree of translational movement loss from orbital implant to ocular prosthesis and analysis will include comparisons between hydroxyapatite and acrylic implants and in patients without an orbital implant, also known as post-enucleation socket syndrome (PESS). A part of this study will also evaluate the accuracy of the two softwares Image J as well as the mediGrid smartphone app in measuring prosthesis motility by comparing it to the ruler as a "gold" standard.

ELIGIBILITY:
Inclusion Criteria:

* Adults with surgery to remove one eye
* Able to give consent and understand the study
* Able to cooperate by following instructions (keeping head still, perform gaze movements)
* Enucleation was performed with the integrated implant technique (recti muscles sutured directly to the scleral cap or the mesh around the implant in a location corresponding to muscle insertion.

Exclusion Criteria:

* Radiotherapy to socket
* Chemotherapy
* Implant exposure repair
* Secondary orbital implant
* Concurrent socket pathology:
* Socket infection
* Socket exposure
* Giant papillary conjunctivitis
* Presence of ocular motility disorders on either side of the face, such as nystagmus, known muscle restrictive disorders (thyroid eye disease, previous trauma, idiopathic orbital inflammatory disease) and neurological disorders (cranial neuropathies, multiple sclerosis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2019-07-18 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
Measurements of orbital implant and ocular prosthesis motility via the mediGrid app | 1 Month
  Orbital implant motility in patient with enucleated sockets will be measured with a mediGrid app. The app will evaluate the degree of translational movement loss from orbital implant to ocular prosthesis.

CONTACTS AND LOCATIONS:
Overall Officials: Mandeep Sagoo, Principal Investigator — Moorfields Eye Hospital NHS Foundation Trust
Locations (1):
- Moorfields Eye Hospital NHS Foundation Trust, 162 City Road, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
All participant data will remain within the sponsor organisation.